CLINICAL TRIAL: NCT06570681
Title: Video Call Assisted Assessment of Acute Stroke in Addition to Stroke Scales in a Prehospital Setting: A Cluster Randomised Controlled Trial
Brief Title: Video Call Assisted Assessment of Acute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHS-Neuro-1-2024
Record Dates: First submitted 2024-05-28; First posted 2024-08-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): If the patient is eligible for study inclusion, eight symptoms from the study protocol are evaluated and registered in the Prehospital Patient Journal (PPJ) on the amPHITM Prehospital Health Care Record (Amphi Systems, Hasserisvej 125, 9000 Aalborg, Denmark), on a tablet mounted in each EMT vehicle. If the vehicle is in the control arm the patient is triaged by the on-call neurologist based on a standard telephone call
- Video call assisted assessment of acute stroke (Active Comparator): If the patient is eligible for study inclusion, the last symptoms from the study protocol are evaluated and registered in the Prehospital Patient Journal (PPJ) on the amPHITM Prehospital Health Care Record (Amphi Systems, Hasserisvej 125, 9000 Aalborg, Denmark), on a tablet mounted in each EMT vehicle. Afterwards the EMS personnel will contact the on-call neurologist and if the vehicle is in the intervention arm a live video stream is initiated. The on-call neurologist then examines the patient via the video-call and triage the patient.
  Interventions: Diagnostic Test: Video call assisted assessment of acute stroke

INTERVENTIONS:
Diagnostic Test: Video call assisted assessment of acute stroke — If the patient is eligible for study inclusion, eight symptoms from the study protocol are evaluated and registered in the Prehospital Patient Journal (PPJ) on the amPHITM Prehospital Health Care Record (Amphi Systems, Hasserisvej 125, 9000 Aalborg, Denmark), on a tablet mounted in each EMT vehicle. Afterwards, the EMS personnel will contact the on-call neurologist and if the vehicle is in the intervention arm a live video stream is initiated. The on-call neurologist then examines the patient via via the video-call and triages the patient.
  Arms: Video call assisted assessment of acute stroke

SUMMARY:
This study aims to investigate whether a live stream video between the on-call neurologist and the emergency medical technicians can increase feasibility and performance of symptom-based prehospital stroke scales.

DETAILED DESCRIPTION:
Treatment of stroke with either thrombolysis or thrombectomy is highly time-dependent (administration within 4.5 hours and 24 hours from symptom onset, respectively), and morbidity and mortality increase with time from symptom onset to treatment. Hence, prehospital evaluation and transport must be as accurate and rapid as possible in order to minimise time to treatment.

Different triage and transport paradigms for patients with suspected stroke are being investigated and multiple stroke scales have been coined in order to examine patients suspected of stroke in a prehospital setting. However, performance and feasibility vary greatly in different validation studies suggesting that those outcomes are greatly dependent on other factors i.e. acceptance amongst stakeholders, implementation process, patient segment etc. Some recent studies have shown promising results using video solutions between emergency medical services (EMS) personnel and on-call neurologist in examining patients suspected of stroke in the prehospital phase. The investigators will perform this trial to examine whether a video call assisted assessment of patients suspected of stroke in a prehospital setting can increase feasibility and performance of symptom-based prehospital stroke scales.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke within 24 hours from onset (confirmed with Prehospital Stroke 1 decision tool)
* Age >18 years

Exclusion Criteria:

* Suspected stroke more than 24 hours ago
* In-hospital stroke or private transport to hospital
* Unconsciousness defined as Glasgow Coma Score (GCS) ≤ 8 (as they cannot be rated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Acute ischemic stroke (AIS) or transient ischemic attack (TIA) diagnosis at discharge | At discharge, assessed within one week from symptom onset
  AIS or TIA as diagnosis. (binary outcome)

SECONDARY OUTCOMES:
Number of patients with acute ischemic stroke (AIS) with LVO on neuroimaging | Within 48 hours of admission
  AIS with LVO on neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography). LVO is defined as a occlusion or sub-occlusion of the intracranial internal carotid artery, middle cerebral artery M1 or M2, basilar artery. Sign of dense cerebral artery on CT is also considered LVO positive. (binary outcome).
Number of patients with Other large vessel AIS | at admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with AIS with occlusion or sub-occlusion of either anterior cerebral artery A1 or A2, posterior cortical artery P1 or intracranial vertebral artery (binary outcome).
Number of patients with verified acute ischemic stroke (AIS) on neuroimaging | Within 48 hours of admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with AIS
Number of patients with Haemorrhagic stroke | at admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with intra cranial haemorrhage (ICH) (binary outcome)

OTHER OUTCOMES:
Duration of examination on video-call | up to 120 minutes prior to admission (prehospital phase)
  Duration of examination on video-call measured in minutes (continuous outcome)
Number of patients which have mimic mistaken for stroke | Through study completion, approximately 2 months
  Mimic mistaken for stroke evaluated as discrepancy between stroke as tentative diagnoses at primary contact from EMS and final diagnosis at discharge
Prehospital time on scene | up to 120 minutes prior to admission (prehospital phase)
  Time on scene from arrival EMS to departure EMS measured in minutes (continuous outcome)
Type of department patient is admitted to after consultation with the neurologist | At admission
  Where was the patient sent after telephone/video consultation with the on-call neurologist.
Door-in-door-out (DIDO) time | at admission
  DIDO times for patients subsequently sent to comprehensive stroke unit for thrombectomy treatment.
Door-to-needle (DNT) time | at admission
  DNT times for patients receiving thrombolysis
Door-to-Groin-Puncture (DTGP) time | within 24 hours of admission
  DTGP times for patients receiving treatment with thrombectomy
Onset-to-Groin-Puncture (OTP) time | within 24 hours of admission
  OTP for patients receiving treatment with thrombectomy
90 days modified Ranking Scale (mRS) | 90 days post admission date
  Modified Rankin Scale score in stroke patients as evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Aabenraa, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No